CLINICAL TRIAL: NCT05862506
Title: Effects of the Daily Mile Program on Health - Related Physical Fitness and Sleep Quality in Overweight/Obese Schoolchildren: a Non- Randomized Clinical Trial
Brief Title: Effects of the Daily Mile Program on General Health in Overweight/Obese Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unidades Tecnológicas de Santander (Other)
Collaborators: Universidad Industrial de Santander (Other)
Responsible Party: Principal Investigator, Adrian Marcel De La Rosa Gonzalez, Doctor, Unidades Tecnológicas de Santander
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BI - 404
Record Dates: First submitted 2023-03-05; First posted 2023-05-17 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Overweight Adolescents; Obesity, Adolescent
Keywords: physical activity; school based program; physical fitness
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Daily Mile (Experimental): The intervention consisted of walking, jogging or running for ~ 15 min (~ one mile) of exercise at a pace self-selected by each individual child, outside the school buildings during recess time, three times a week during 10 weeks. Children were instructed to maintain active for the full 15 min and, if necessary, to stop for resting only occasionally.
  Interventions: Behavioral: Daily Mile
- Control Group (No Intervention): This group will be received only the physical education lessons and it will be followed-up equally to compare outcomes in the future.

INTERVENTIONS:
Behavioral: Daily Mile — The intervention consisted of walking, jogging or running for ~ 15 min (~ one mile) of exercise at a pace self-selected by each individual child, outside the school buildings during recess time, three times a week during 10 weeks. Children were instructed to maintain active for the full 15 min and, if necessary, to stop for resting only occasionally.
  Arms: The Daily Mile

SUMMARY:
This study is a clinical trial will be carried out during academic term to assess the potential effects of the Daily Mile program on health-related physical fitness and sleep quality on overweight/obese schoolchildren.The trial will be taken place in Bucaramanga, Colombia

DETAILED DESCRIPTION:
Introduction: Regular physical activity is essential for promoting health and well-being, especially during childhood and adolescence. The World Health Organization (WHO) recommends that children and adolescents (ages 5 to 17 years) should average 60 minutes of moderate-to-vigorous intensity physical activity per day, primarily of aerobic capacity, with the aim of preventing and/or reducing the incidence of overweight non-communicable diseases in adulthood and modifying emotional behaviors such as enjoyment, intrinsic motivation and perceived autonomy, among others. Modifications in these recommendations have probably been generated due to the increase of physical inactivity prevalence and sedentary behaviours in the population, which have been related to an increased risk of obesity, cardiovascular disease, diabetes, coronary heart disease and stroke, as well as delayed cognitive development and decreased in the academic performance of children and young people.

Recently, the WHO classified physical inactivity as the fourth mortality risk factor with 6%, after hypertension (13%), smoking (9%) and diabetes (6%)9. In Colombia, the National Survey of the Nutritional Situation (ENSIN 2015) found that only 35.8% of boys and 26% of girls between 6 and 12 years of age complied with the physical activity recommendations.

The previous Survey shows that 25.3% of boys and 23.5% of girls between 5 and 12 years of age are overweight or obese, which means an increase of 5.1%. and 6.2% respectively in relation to the year 2010 and 10.1% and 9.8% in relation to the year 2005, indicating a substantial increase in the data related to body weight In Colombia. In 2016 worldwide, it was estimated that the number of children under five years of age with obesity exceeded 41 million. In the same way, it has been found that the presence of overweight and obesity increases the probability of the development of non-communicable diseases such as diabetes, cardiovascular diseases and metabolic syndromes.

In response to this situation, one of the objectives established by the WHO's global action plan on physical activity 2018-2030 was to reduce the prevalence of physical inactivity by 10% by 2025 and 15% by 2030. For this reason, two of the strategic objectives have been called "Create active environments" and "create active people", whose purpose is to create and promote spaces and access to programs and opportunities that increase physical activity in their different communities and, that in the case of the school population, a greater participation in physical activity leads to a greater capacity for concentration and cognitive function, which could result in an improvement in academic performance.

A physical activity program to be developed in school environments is The Daily Mile (DM). It is an initiative created at St Ninian Primary School (Stirling, Scotland) in 2012 that was initially proposed as a solution to a perceived lack of physical fitness in children between 5 and 12 years of age. The DMaily Mile encompasses a 15-minute walking, jogging or running each day, without additional material resources or clothing, within their class time.

Although the Daily Mile program has grown in popularity among schools in the United Kingdom, the United States, Italy, and the Netherlands, among others, there is no evidence of research carried out on schoolchildren implementing this program in Colombia or in overweight/obese children. There is an urgent need for results from well-designed experimental studies that enable a better understanding of the impact of exercise in school environments on various health outcomes.

Methodology: The intervention will start in the middle of the first academic term. The Daily Mile intervention will be consisted of walking, jogging or running for ~ 15 min (~ one mile) of exercise at a pace self-selected by each individual child, outside the school buildings during recess time, three times a week. Children were instructed to maintain active for the full 15 min and, if necessary, to stop for resting only occasionally. The program will be guided and supervised by physical education professionals previously trained. All the sessions will take place at the outside School buildings.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled at the school.
* Be aged between 11 and 17 years, healthy (physically, psychologically and cognitively).
* Present a BMI greater than or equal to the 85th percentile for their gender and age, according to WHO (World Health Organization).
* Be free of any medication that could interact with the protocol (e.g., cardiac abnormalities, hypertension, diabetes, orthopaedic, neuromuscular, or neurological disorders).
* Present no contraindication to physical activity

Exclusion Criteria:

- Perform any scheduled physical activity outside the curricula.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity | At the end of the intervention period (10 weeks)
  maximum oxygen consumption in ml/kg*min, distance covered in meters

SECONDARY OUTCOMES:
Muscle strength | At the end of the intervention period (10 weeks)
  in Newtons
Body composition | At the end of the intervention period (10 weeks)
  In fat and muscle mass kilograms
Cardiometabolic biomarkers | At the end of the intervention period (10 weeks)
  glucose and lipid profile in mg/dL
Physical activity level | At the end of the intervention period (10 weeks)
  in minutes per week
Sleep quality | At the end of the intervention period (10 weeks)
  Pittsburgh Sleep Quality Index, provides an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidades tecnológicas de Santander, Bucaramanga, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breheny K, Passmore S, Adab P, Martin J, Hemming K, Lancashire ER, Frew E. Effectiveness and cost-effectiveness of The Daily Mile on childhood weight outcomes and wellbeing: a cluster randomised controlled trial. Int J Obes (Lond). 2020 Apr;44(4):812-822. doi: 10.1038/s41366-019-0511-0. Epub 2020 Jan 28. PMID 31988481
- [Background] Chesham RA, Booth JN, Sweeney EL, Ryde GC, Gorely T, Brooks NE, Moran CN. The Daily Mile makes primary school children more active, less sedentary and improves their fitness and body composition: a quasi-experimental pilot study. BMC Med. 2018 May 10;16(1):64. doi: 10.1186/s12916-018-1049-z. PMID 29743076
- [Background] Brustio PR, Mulasso A, Marasso D, Ruffa C, Ballatore A, Moise P, Lupo C, Rainoldi A, Boccia G. The Daily Mile: 15 Minutes Running Improves the Physical Fitness of Italian Primary School Children. Int J Environ Res Public Health. 2019 Oct 15;16(20):3921. doi: 10.3390/ijerph16203921. PMID 31618975